CLINICAL TRIAL: NCT04908709
Title: Spectroscopic MRI Guided Proton Therapy for Pediatric High-Grade Glioma (RAD4500)
Brief Title: Spectroscopic MRI Guided Proton Therapy in Assessing Metabolic Change in Pediatric Patients With Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bree Eaton, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106849; NCI-2018-02065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00106849; RAD4500-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-05-20; First posted 2021-06-01 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Malignant Brain Glioma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Diagnostic (sMRI) (Experimental): Patients undergo sMRI over less than 1 hour within 7 days prior to start of standard of care radiation therapy and at 10 weeks.
  Interventions: Procedure: Magnetic Resonance Spectroscopic Imaging; Device: Proton Therapy
- Group 2 (Active Comparator): Patients will undergo 3-4 sMRI scans at baseline prior to RT, 1 month, 4 months, and 7 months after RT, and/or at any time of suspected tumor recurrence.
  Interventions: Procedure: Magnetic Resonance Spectroscopic Imaging; Device: Proton Therapy

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo sMRI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging
Device: Proton Therapy — Target volume treatment
  Other Names: Spectroscopic MRI; Proton Radiation Therapy; sMRI imaging; Magnetic Resonance Spectroscopy; 3D whole brain MR spectroscopic imaging sequence

SUMMARY:
This trial studies how well spectroscopic magnetic resonance imaging (MRI) guided proton therapy works in assessing metabolic change in pediatric patients with brain tumors. The non-invasive imaging, such as spectroscopic MRI may help to map the differences in tumor metabolism compared to healthy tissue without injection of any contrast agent.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain spectroscopic (s)MRI data from pediatric high grade glioma (HGG) patients before receiving standard of care radiation therapy (RT) and correlate baseline Cho/NAA ratios to recurrence patterns. (Cohort 1, observational) II. To assess the feasibility and safety of using sMRI to define proton therapy high dose (60Gy) target volumes for treatment delivery. (Cohort 2, intervention)

SECONDARY OBJECTIVES:

I. To evaluate how Cho/NAA defined radiation target volumes compare to standard of care radiation target volumes in size and resulting radiation delivery to adjacent normal tissue, by creating mock comparison RT plans for each patient.

II. To compare voxel-to-voxel changes in pre-treatment and post-treatment sMRI and evaluate as potential early predictor of tumor response/recurrence.

III. To evaluate sMRI as a tool in identifying pseudoprogression vs. true progression and correlate post-treatment sMRI metabolite ratios with histopathology if collected.

IV. To report patterns of failure in relationship to the RT field (local, marginal, or distant), progression-free survival (PFS) and overall survival (OS) among all patients.

V. To report patient reported outcomes of health related quality of life (QOL) during and after proton therapy for pediatric HGG.

VI. To build a longitudinal tracking database including clinical data, imaging, and genomic molecular profiling for pediatric HGG treatment.

OUTLINE:

Patients undergo sMRI prior to radiation therapy, at 1, 4, and 7 months after RT, and at the time of suspected recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed high-grade glioma (World Health Organization [WHO] grade 3-4). Patients with a radiographically diagnosed high-grade glioma may enroll prior to pathologic confirmation, but would be removed from study if pathology did not confirm the diagnosis of high-grade glioma.
* Primary tumor located within the supratentorial brain.
* Recommended to receive definitive radiation therapy.
* Able to receive MRI scans.
* Both males and females, and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients with pacemakers, non-titanium aneurysm clips, neurostimulators, cochlear implants, non-titanium metal in ocular structures, or other incompatible implants which makes MRI safety an issue are excluded.
* Patients that have any significant medical illnesses that in the investigator's opinion cannot be adequately tolerate MRI scan are excluded.
* Pathology demonstrated low-grade glioma or other benign or non-invasive brain tumor.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2029-10-13 (Estimated); Study Completion 2030-10-13 (Estimated)

PRIMARY OUTCOMES:
Cho/NAA ratios at baseline in tumor and in regions of tumor recurrence in patients receiving standard of care radiotherapy | Through study completion, an average of 1 year
  The spatial relationship between baseline sMRI abnormalities and tumor recurrence will be reported and proportion of overlap will be quantified.
Incidence of adverse events | Through study completion, an average of 1 year
  Toxicity will be defined according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Feasibility of using sMRI to define proton therapy high dose (60Gy) target volumes for treatment delivery | From Baseline up to 3 years from treatment
  Will be estimated by the Kaplan-Meier Method.

CONTACTS AND LOCATIONS:
Overall Officials: Bree R Eaton, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia